CLINICAL TRIAL: NCT07309289
Title: NALIRIFOX Plus Targeted Therapy Versus FOLFOX Plus Targeted Therapy as First-line Treatment for Metastatic Colorectal Cancer: a Multicentre, Open-label, Randomised Trial
Brief Title: NALIRIFOX Plus Targeted Therapy Versus FOLFOX Plus Targeted Therapy as First-line Treatment for Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Tianshu Liu, Director, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DEY-CRC-K10
Record Dates: First submitted 2025-12-15; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Colorectal Cancer (CRC)
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NALIRIFOX plus targeted therapy (Experimental): NALIRIFOX plus targeted therapy
  Interventions: Drug: NALIRIFOX plus targeted therapy
- FOLFOX plus targeted therapy (Active Comparator): FOLFOX plus targeted therapy
  Interventions: Drug: FOLFOX plus targeted therapy

INTERVENTIONS:
Drug: NALIRIFOX plus targeted therapy — Drug: Irinotecan Liposome Irinotecan liposome injection will be administered by an intravenous infusion at the dose of 50 mg/m^2, d1, 14 days per cycle.
  Drug: Oxaliplatin 75 mg/m^2, intravenously infusion, d1, 14 days per cycle. Drug: 5-FU 2400mg/m^2, intravenous infusion, d1-2, 14 days per cycle. Drug: LV/l-LV 400mg/m^2 or 200mg/m^2 , intravenous infusion, d1, 14 days per cycle. Drug: Bevacizumab 5mg/kg, intravenous infusion, d1, 14 days per cycle. Drug: Cetuximab 500mg/m^2, intravenous infusion, d1, 14 days per cycle.
  Arms: NALIRIFOX plus targeted therapy
Drug: FOLFOX plus targeted therapy — Drug: Oxaliplatin 85 mg/m^2, intravenously infusion, d1, 14 days per cycle. Drug: 5-FU 2400mg/m^2, intravenous infusion, d1-2, 14 days per cycle. Drug: LV/l-LV 400mg/m^2 or 200mg/m^2 , intravenous infusion, d1, 14 days per cycle. Drug: Bevacizumab 5mg/kg, intravenous infusion, d1, 14 days per cycle. Drug: Cetuximab 500mg/m^2, intravenous infusion, d1, 14 days per cycle.
  Arms: FOLFOX plus targeted therapy

SUMMARY:
To explore the safety and efficacy of NALIRIFOX plus targeted therapy versus FOLFOX plus targeted therapy as first-line treatment for metastatic colorectal cancer.

DETAILED DESCRIPTION:
This is a multicentre, open-label, randomised study to explore the safety and efficacy of NALIRIFOX plus targeted therapy versus FOLFOX plus targeted therapy as first-line treatment for metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Histopathologically confirmed patient with an inoperable metastatic colorectal adenocarcinoma
* The unresectable stage of metastatic disease has not received any systemic antitumor therapy
* For subjects previously receiving neoadjuvant or adjuvant therapy, the date of first discovery of disease progression must be at least 12 months removed from the date of last administration of neoadjuvant or adjuvant therapy
* The presence of at least 1 measurable lesion that can be evaluated according to the RECIST v1.1 criteria
* ECOG 0~1
* Normal bone marrow and organ function
* Understand the situation of this study, patients and/or legal representatives voluntarily agree to participate in this study and sign informed consent form

Exclusion Criteria:

* Patients with known MSI-H or dMMR who were evaluated by investigators as suitable for treatment with immune checkpoint inhibitors.
* Patients allergic to the investigational drug and its excipients
* Underweight (body mass index [BMI]<18.5 kg/m^2
* Known or suspected central nervous system metastasis
* Received irinotecan before enrollment
* Had undergone surgery and other oncologic treatments within the first 4 weeks of enrollment
* Previous treatment-related toxicity didn't return to NCI-CTCAE v5.0 class I or below.
* The use of CYP3A, CYP2C8, and UGT1A1 inhibitors or inducers couldn't be discontinued or were not discontinued within 2 weeks prior to enrollment
* Serious gastrointestinal disorders
* Interstitial lung disease
* Tendency of arterial embolism and massive bleeding within 6 months before enrollment (except surgical bleeding)
* Patients with fluid accumulation that couldn't reach a stable state and small amount of pleural effusion or ascites on imaging without clinical symptoms could be enrolled
* Intestinal obstruction, or a risk of intestinal obstruction in the short term
* Gastrointestinal perforation, intraperitoneal abscess, and fistula
* Any serious or uncontrolled systemic disease, including uncontrolled high blood pressure, heart disease, active bleeding, active viral infection, etc
* Have had other malignancies within the past 5 years or currently, except cured cervical carcinoma in situ, uterine carcinoma in situ, and non-melanoma skin cancer
* Patients of childbearing age who refuse to take contraceptives, women who are pregnant or breastfeeding
* The researchers didn't consider it appropriate to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
18 month PFS rate | Eighteen months after the randomization of research participants
  To investigate the preliminary antitumor efficacy of study.

SECONDARY OUTCOMES:
Objective response rate | From date of randomization until the date of first documented progression、termination of treatment, or date of death from any cause, whichever came first, assessed up to 12 months
  To investigate the preliminary antitumor efficacy of study.
Disease control rate | From date of randomization until the date of first documented progression、termination of treatment, or date of death from any cause, whichever came first, assessed up to 12 months
  To investigate the preliminary antitumor efficacy of study.
Progression free survival | From date of randomization until the date of first documented progression、termination of treatment, or date of death from any cause, whichever came first, assessed up to 12months
  To investigate the preliminary antitumor efficacy of study.
R0 resection | From date of randomization until the date of surgical resection, assessed up to 12 months
  To assess surgical conversion rates in patients who could be surgically resected.
Overall survival | From date of randomization until the date of death from any cause, assessed up to 30 months
  To investigate the preliminary antitumor efficacy of study.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, China